CLINICAL TRIAL: NCT06928792
Title: Effects Of Quadratus Lumborum Release on Respiratory Outcomes on Low Back Pain Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/02134 Suleman
Record Dates: First submitted 2025-02-20; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Low Back Pain
Keywords: Respiratory function test; Numeric Pain rating scale; METs; Chronic pain
MeSH Terms: conditions — Low Back Pain; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to the experimental group or control group after a baseline assessment with a lottery ticket and an opaque envelope containing the same number of folded papers labeled "control" or "intervention." Each participant took a piece of paper that identified their group and gave it to the researchers without seeing what was written. Participants were not notified which group was assigned.
Who Masked: Participant, Outcomes Assessor
Masking Description: The researchers who evaluated the participants were not informed of how the participants were grouped. Participants were informed that they would receive one of two different interventions without indicating which group should undergo METs on Quadratus lumborum or Conventional treatment for chronic low back pain.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: interventional group A: Muscle Energy Technique (MET) (Experimental): 10 min hot pack application, followed by MET on the Quadratus Lumborum (3 reps with a 7s hold). Flexibility exercises include William flexion with b/L knee-to-chest stretches (10s hold, repeated 10 times) and static stretching of the hamstrings, gastrocnemius, and IT band (5 reps, 5s hold). Strengthening exercises comprise isometric hip flexor activation (5 reps with a 15s hold), side planks (3 reps, 30s hold), and static side bending (5 reps, 10s hold). The intervention will be performed once daily, consisting of 3 sets per session, continued for 4 weeks to enhance flexibility, core stability, and muscular balance, ultimately contributing to pain relief and improved functional mobility in CLBP patients
  Interventions: Other: Experimental interventional group A, (MET).
- Control :interventional group B: (conventional intervention exercises) (Active Comparator): 10-minute hot pack application, followed by William flexion with bilateral knee-to-chest stretches (10s hold, reps 10 times). Flexibility exercises consist of static stretching for the hamstrings, gastrocnemius, and iliotibial band (5 reps with a 5s hold). Strengthening exercises include isometric hip flexor activation (5 reps with a 15s hold), side planks (3 reps with a 30s hold), and static side bending (5 reps with a 10s hold). The protocol will be performed once daily, with 3 sets per session, continued for 4 weeks to improve flexibility, core stability, and pain management in CLBP patients.
  Interventions: Other: Control: group B (conventional intervention exercises)

INTERVENTIONS:
Other: Experimental interventional group A, (MET). — 10-minute hot pack application, followed by MET on the Quadratus Lumborum (3 repetitions with a 7-second hold). Flexibility exercises include William flexion with bilateral knee-to-chest stretches (10-second hold, repeated 10 times) and static stretching of the hamstrings, gastrocnemius, and iliotibial band (5 repetitions with a 5-second hold). Strengthening exercises comprise isometric hip flexor activation (5 repetitions with a 15-second hold), side planks (3 repetitions with a 30-second hold), and static side bending (5 repetitions with a 10-second hold). The intervention will be performed once daily, consisting of 3 sets per session, continued for 4 weeks to enhance flexibility, core stability, and muscular balance, ultimately contributing to pain relief and improved functional mobility in CLBP patients
  Arms: Experimental: interventional group A: Muscle Energy Technique (MET)
Other: Control: group B (conventional intervention exercises) — 10-minute hot pack application, followed by William flexion with bilateral knee-to-chest stretches (10-second hold, repeated 10 times). Flexibility exercises consist of static stretching for the hamstrings, gastrocnemius, and iliotibial band (5 repetitions with a 5-second hold). Strengthening exercises include isometric hip flexor activation (5 repetitions with a 15-second hold), side planks (3 repetitions with a 30-second hold), and static side bending (5 repetitions with a 10-second hold). The protocol will be performed once daily, with 3 sets per session, continued for 4 weeks to improve flexibility, core stability, and pain management in CLBP patients.
  Arms: Control :interventional group B: (conventional intervention exercises)

SUMMARY:
The aim of this research is to check the effects of Quadratus Lumborum (QL) release on respiratory function and pain levels in individuals with chronic low back pain. Randomized controlled trials done at Pakistan Railway General Hospital, Rawalpindi and Rawal General & Dental Hospital Islamabad. The sample size was 36. The subjects were divided into two groups, 18 subjects in the experimental group will receive muscle energy technique on quadratus lumborum along with conventional intervention for LBP and 18 in control group will only receive conventional intervention exercises for LBP. Study duration was of 6 months. Sampling technique applied was non probability connivance sampling technique. Only 30-60 years both males and females diagnosed with mechanical low back pain persist at least >3 months. Tools used in the study of Numeric Pain rating scale (Pain assessment). Modified Oswestry Disability Index (m-ODI) (for ADLs in CLBP). Inclinometer (for ranges of lumber spine). Digital spirometer (for FEV1/FVC ratio). Inches Tap (For Chest Expansion) & (For Quadratus lumborum length test). Fatigue Severity Scale (FSS).

DETAILED DESCRIPTION:
The aim of this research is to check the effects of Quadratus Lumborum (QL) release on respiratory function and pain levels in individuals with chronic low back pain. Randomized controlled trials done at Pakistan Railway General Hospital, Rawalpindi and Rawal General & Dental Hospital Islamabad. The sample size was 36. The subjects were divided into two groups, 18 subjects in the experimental group will receive muscle energy technique on quadratus lumborum along with conventional intervention for LBP and 18 in control group will only receive conventional intervention exercises for LBP. Study duration was of 6 months. Sampling technique applied was non probability connivance sampling technique. Only 30-60 years both males and females diagnosed with mechanical low back pain persist at least >3 months. Tools used in the study of Numeric Pain rating scale (Pain assessment). Modified Oswestry Disability Index (m-ODI) (for ADLs in CLBP). Inclinometer (for ranges of lumber spine). Digital spirometer (for FEV1/FVC ratio). Inches Tap (For Chest Expansion) & (For Quadratus lumborum length test). Fatigue Severity Scale (FSS).

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-60 years.
2. Both Genders: Male and Female.
3. Diagnosed with mechanical low back pain persist at least >3 months.
4. Self-evaluation of the breathing questionnaire, SEBQ >11.
5. The patient exhibits decreased pulmonary functional volumes compared to the normal values, which include FEV, FVC,FEV₁/FVC
6. The Quadratus Lumborum length test in side-lying inches indicates QL shortening.
7. Patient with either unilateral or bilateral Quadratus lumborum tightness but intervention will be given on both sides.
8. Numeric Pain Rating > 3/10.

Exclusion Criteria:

1. Diagnosed chronic respiratory disease (e.g., asthma, COPD, bronchitis).
2. Diagnosed non-mechanical low back pain (e.g., ankylosing spondylitis, tumors).
3. Diagnosed lumbar spine surgery within the last 12 months.
4. Diagnosed significant neurological deficits.
5. Spinal injuries or other comorbidities.
6. Infection, trauma, pregnancy, fracture, or fall.
7. Unable to understand and follow the commands.
8. Unwillingness to comply with the follow-up schedule.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-07 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain rating scale. | baseline measurement to 2 weeks
  It is the tool to measure pain intensity It ranges from 0 to 10. If the patient feels no pain, then 0 will be marked. 5 shows moderate pain and 10 will be marked if pain is most extreme ever felt by the patient.(10) The patients were asked to mark the point they felt their pain accordingly
Digital spirometer. | baseline measurement to 2 weeks
  Spirometry is a vital pulmonary function test used to assess lung health by measuring Peak Expiratory Flow (PEF)
Inches Tap (For Chest Expansion) | baseline measurement to 2 weeks after every session.
  Chest expansion was measured in a standing position with elbows slightly flexed and hands on hips, using a non-stretchable inch tape at the 2nd intercostal space (ICS), 4th ICS, and xiphoid process. Participants performed maximal deep inspiration and expiration, and the difference was recorded.
Fatigue Severity Scale (FSS) | baseline measurement to 2 weeks.
  Unidimensional, nine-item self-reported questionnaire designed to assess the severity and impact of fatigue on daily functioning and quality of life over the past week. Participants rate each item on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree), with higher scores indicating greater fatigue severity. The total score is calculated by summing the individual item scores, resulting in a range from 9 to 63, with a score of ≥36 indicating significant fatigue.

SECONDARY OUTCOMES:
Inclinometer for Lumbar Flexion. | baseline measurement to 2 weeks after every session
  The inclinometer is a reliable and valid tool for measuring lumbar range of motion (ROM), including flexion, extension, and side bending. To use the inclinometer, place one device on the T12 vertebra and another on the S1 vertebra while the patient stands in a neutral posture. The patient then performs forward bending.
Inclinometer for Lumbar Extension. | baseline measurement to 2 weeks after every session
  The inclinometer is a reliable and valid tool for measuring lumbar range of motion (ROM), including flexion, extension, and side bending. To use the inclinometer, place one device on the T12 vertebra and another on the S1 vertebra while the patient stands in a neutral posture. The patient then performs lumbar extension.
Inclinometer for Lumbar Side Bending (Rt) | baseline measurement to 2 weeks after every session
  The inclinometer is a reliable and valid tool for measuring lumbar range of motion (ROM), including flexion, extension, and side bending. To use the inclinometer, place one device on the T12 vertebra and another on the S1 vertebra while the patient stands in a neutral posture. The patient then performs movements for right-side bending.
Inclinometer for Lumbar Side Bending (Lt) | baseline measurement to 2 weeks after every session
  The inclinometer is a reliable and valid tool for measuring lumbar range of motion (ROM), including flexion, extension, and side bending. To use the inclinometer, place one device on the T12 vertebra and another on the S1 vertebra while the patient stands in a neutral posture. The patient then performs left-side bending.
Inclinometer for Lumbar Rotation (Rt) | baseline measurement to 2 weeks after every session
  The inclinometer is a reliable and valid tool for measuring lumbar range of motion (ROM), including flexion, extension, and side bending. To use the inclinometer, place one device on the T12 vertebra and another on the S1 vertebra while the patient stands in a neutral posture. The patient then performs right rotation at lumbar
Inclinometer for Lumbar Rotation (Lt) | baseline measurement to 2 weeks after every session
  The inclinometer is a reliable and valid tool for measuring lumbar range of motion (ROM), including flexion, extension, and side bending. To use the inclinometer, place one device on the T12 vertebra and another on the S1 vertebra while the patient stands in a neutral posture.The patient then performs Left rotation at lumbar.

CONTACTS AND LOCATIONS:
Overall Officials: Aisha Razzaq, PHD*, Principal Investigator — Riphah International University
Locations (1):
- Rawal Institute of Rehabilitation Sciences, Islamabad, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No